CLINICAL TRIAL: NCT04551911
Title: A Randomized, Double-Blind Placebo-Controlled Study to Evaluate the Safety and Efficacy of Rayaldee (Calcifediol) Extended-release Capsules to Treat Symptomatic Patients Infected With SARS-CoV-2 (REsCue)
Brief Title: Safety and Efficacy of Rayaldee for Treating Mild to Moderate COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTAP101-CL-2014
Record Dates: First submitted 2020-09-15; First posted 2020-09-16 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: COVID-19; Coronavirus; SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Calcifediol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rayaldee (Experimental): Subjects will be instructed to take a loading dose of 10 capsules (300 mcg) of study drug per day on Days 1, 2 and 3 at bedtime after fasting for at least 3 hours following dinner, with any nonalcoholic liquid, by the oral route. On Days 4-27, subjects will take a maintenance dose of 2 capsules per day at bedtime unless otherwise directed. Patients were to remain fasted for at least 3 hours after administration of study drug.
  Interventions: Drug: Rayaldee
- Placebo (Placebo Comparator): Subjects will be instructed to take a loading dose of 10 capsules (0 mcg) of study drug per day on Days 1, 2 and 3 at bedtime after fasting for at least 3 hours following dinner, with any nonalcoholic liquid, by the oral route. On Days 4-27, subjects will take a maintenance dose of 2 capsules per day at bedtime unless otherwise directed. Patients were to remain fasted for at least 3 hours after administration of study drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rayaldee — 30 mcg calcifediol Extended-Release (ER) Capsule
  Other Names: CTAP101 Capsule
  Arms: Rayaldee
Drug: Placebo — 0 mcg calcifediol Extended-Release (ER) Capsule
  Arms: Placebo

SUMMARY:
This is a phase 2, single or multi-center, randomized, double-blind placebo-controlled study to evaluate the safety and efficacy of Rayaldee (CTAP101 Capsules) to treat adult subjects with mild to moderate COVID-19 who test positive for SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age
2. Confirmed within the past 3 days to have SARS-CoV-2 infection as evidenced by a positive nasopharyngeal swab test using RT-PCR or any substitutable FDA-authorized diagnostic test
3. Confirmed to have only mild or moderate COVID-19 based on the first of the patient reported scores obtained during screening which meets the criterion a FLU-PRO Plus© score of ≥ 1.5 for each of the chest/respiratory and body/systemic domains, and the absence of clinical signs indicative of more severe disease (eg, oxygen saturation < 94% on room air or respiration rate > 30 bpm)
4. Represents on self-assessment that the current COVID-19 symptoms are not consistent with usual health and that they are the same or worse than on the previous day
5. Willing to limit the use of vitamin D therapies or supplements except for normally fortified food products (eg, milk) during the course of the 6-week study
6. Must demonstrate the ability to comply with all study requirements
7. Must be without any disease state or physical condition that might impair evaluation of safety or which, in the investigator's opinion, would interfere with study participation.

Exclusion Criteria:

1. Clinical signs indicative of severe or critical COVID-19 disease (eg, oxygen saturation < 94% on room air or respiration rate > 30 bpm)
2. Pregnant or lactating women who are breastfeeding
3. Use of systemic glucocorticoid medications in the last six months
4. Recent history (previous 12 months) of primary hyperparathyroidism, kidney stones, hypercalciuria and/or hypercalcemia
5. History of a chronic granuloma-forming disease (eg, sarcoidosis)
6. History of tuberculosis or histoplasmosis
7. History of chronic liver disease
8. History (previous 12 months) of cardiac event indicative of chronic cardiovascular diseases including congestive heart failure, poorly controlled hypertension and arrhythmias
9. History in the past five years of multiple myeloma or carcinoma of the breast, lung or prostate
10. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of vitamin D or 25-hydroxyvitamin D (25D) (eg, small bowel resection, history of Crohn's disease or ulcerative colitis)
11. Ongoing treatment with thiazide diuretics
12. History of hyperphosphatemia, hyperuricemia and gout
13. Renal impairment measured as eGFR< 15 mL/min/1.73m² on serum creatinine in the last three months
14. Serum calcium ≥9.8 mg/dL in the last three months
15. Evidence of existing or impending dehydration
16. Known or suspected to have hypersensitivity to any of the constituents of the study drug
17. Currently participating in, or have participated in, an interventional/investigational study within 30 days prior to study screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akhtar Ashfaq, MD FACP FASN, Study Director — OPKO Health, Inc.
Locations (9):
- United States (9):
  - OPKO Investigative Site, San Francisco, California
  - OPKO Investigative Site, Miami, Florida
  - OPKO Investigative Site, Evanston, Illinois
  - OPKO Investigative Site, Laurel, Maryland
  - OPKO Investigative Site, Farmington Hills, Michigan
  - OPKO Investigative Site, Jackson, Michigan
  - OPKO Investigative Site, Sterling Heights, Michigan
  - OPKO Investigative Site, Brookhaven, Mississippi
  - OPKO Investigative Site, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Rayaldee: Subjects will be instructed to take a loading dose of 10 capsules (300 mcg) of study drug per day on Days 1, 2 and 3 at bedtime after fasting for at least 3 hours following dinner, with any nonalcoholic liquid, by the oral route. On Days 4-27, subjects will take a maintenance dose of 2 capsules per day at bedtime unless otherwise directed. Patients were to remain fasted for at least 3 hours after administration of study drug.
  Rayaldee: 30 mcg Extended-Release (ER) Capsule
- Placebo: Subjects will be instructed to take a loading dose of 10 capsules (0 mcg) of study drug per day on Days 1, 2 and 3 at bedtime after fasting for at least 3 hours following dinner, with any nonalcoholic liquid, by the oral route. On Days 4-27, subjects will take a maintenance dose of 2 capsules per day at bedtime unless otherwise directed. Patients were to remain fasted for at least 3 hours after administration of study drug.
  Placebo: 0 mcg Extended-Release (ER) Capsule
Period: Overall Study
Arm/Group | Rayaldee | Placebo
Started | 85 | 86
Completed | 70 | 71
Not Completed | 15 | 15
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Did not receive the study drug | 3 | 4

BASELINE CHARACTERISTICS:
Population: Analysis is for the per protocol population, subjects who had a baseline aggregate five symptom score of >5 and did not have a major protocol deviation prior to resolution.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rayaldee | Placebo | Total
Number analyzed (Participants) | 65 | 69 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (14.13) | 43.8 (14.32) | 43.0 (14.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 41 | 79
  Male | 27 | 28 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 56 | 111
  Not Hispanic or Latino | 10 | 13 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 58 | 65 | 123
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Height [Mean (Standard Deviation); unit: cm] | 167.91 (9.375) | 167.34 (8.747) | 167.62 (9.027)
Weight [Mean (Standard Deviation); unit: kg] | 81.05 (18.730) | 84.27 (18.985) | 82.71 (18.860)
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.62 (5.521) | 29.99 (5.913) | 29.32 (5.746)
eGFR (glomerular filtration rate) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 97.5 (16.89) | 98.5 (18.62) | 98.0 (17.74)
Serum total 25-hydroxyvitamin D (25D) [Mean (Standard Deviation); unit: ng/mL] | 37.7 (12.15) | 37.1 (15.60) | 37.4 (13.98)
Flu-Pro Plus Aggregate Score [Mean (Standard Deviation); unit: scores on a scale] — The Flu-Pro Plus Aggregate Score is computed as the summation of scores from the five individual COVID-19 symptoms (Trouble Breathing, Chest Congestion, Dry or Hacking Cough, Body Aches or Pains, and Chills or Shivering). Individual symptom scores range from 0 (symptom-free) to 4 (very severe symptoms). The total score range is from 0 to 20.
  scores on a scale | 12.8 (3.84) | 12.5 (3.91) | 12.7 (3.86)

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Serum Total 25-hydroxyvitamin D Attained at or Above 50 ng/mL at Visit 3 (Day 14).
Description: Number and percentage of subjects with serum total 25-hydroxyvitamin D attained at or above 50 ng/mL at Visit 3 (Day 14)
Time Frame: 14 days
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Rayaldee | Placebo
Number analyzed (Participants) | 65 | 69
Participants | 51 | 10

2. Primary Outcome: Resolution of COVID-19 Five Aggregated Symptoms Using the Flu-PRO Plus© Questionnaire.
Description: The FLU- PRO Plus© questionnaire was specifically designed and validated to evaluate in clinical trials the presence, severity and duration of symptoms associated with viral infections. It contains 32 items (eg, felt hot, sweating, headache), grouped into 6 domains, that provide a comprehensive evaluation of such symptoms, using 5-point scales (values ranging from 0 to 4) with higher scores indicating worse symptoms. The number of days to resolution of the selected five COVID-19 symptoms (trouble breathing, chest congestion, dry or hacking cough, body aches and pains, and chills and shivering), defined as a reduction in the aggregate symptom score recorded on Day 0 (prior to study drug initiation) by the FLU-PRO Plus© questionnaire to or below 5 for a minimum of three consecutive days. Flu-PRO Plus© was created and supplied by Dr. John Powers and Leidos Biomedical, and the National Institute for Allergy and Infectious Diseases (NIAID).
Time Frame: 42 days
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rayaldee | Placebo
Number analyzed (Participants) | 65 | 69
days | 9.8 (8.15) | 10.8 (9.54)

3. Secondary Outcome: Time to Resolution of COVID-19 Five Aggregated Symptoms
Description: The number of days to resolution of five symptoms (trouble breathing, chest congestion, dry or hacking cough, body aches and pains, and chills and shivering), as measured by the FLU-PRO Plus© questionnaire, with resolution defined as the first aggregate symptom score of ≤5 which is maintained for a minimum of three consecutive days, with no individual symptom score >1
Time Frame: 42 days
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rayaldee | Placebo
Number analyzed (Participants) | 65 | 69
days | 12.0 (8.70) | 12.6 (9.09)

4. Secondary Outcome: Number of Subjects Who Had an COVID-19 Five Aggregated Symptoms Score >5 at Baseline Who Experienced Symptom Resolution as of Day 10
Description: Resolution, defined as the first score of ≤5 which was maintained for a minimum of three consecutive days (without subsequent relapse), for the aggregate five COVID-19 symptoms (trouble breathing, chest congestion, dry or hacking cough, body aches and pains, and chills and shivering) and for each individual symptom, defined as a score of 0 or 1, as measured by the FLU-PRO Plus© questionnaire as of Day 10
Time Frame: 10 days
Population: Per protocol population
Measure: Number; unit: Number of participants
Arm/Group | Rayaldee | Placebo
Number analyzed (Participants) | 65 | 69
Number of participants | 38 | 41

5. Secondary Outcome: Proportion of Subjects Who Had an COVID-19 Five Aggregated Symptoms Score >5 at Baseline Who Experienced Symptom Resolution as of Day 10
Description: Resolution, defined as the first score of ≤5 which was maintained for a minimum of three consecutive days (without subsequent relapse), for the aggregate five COVID-19 symptoms (trouble breathing, chest congestion, dry or hacking cough, body aches and pains, and chills and shivering) and for each individual symptom, defined as a score of 0 or 1, as measured by the FLU-PRO Plus© questionnaire as of Day 10.
  Logistic regression with treatment as the main effect, and baseline aggregate symptom score, baseline 25D level, and body weight as covariates.
Time Frame: 10 days
Population: Per protocol population
Measure: Number; unit: Proportion
Arm/Group | Rayaldee | Placebo
Number analyzed (Participants) | 65 | 69
Proportion | 0.618 | 0.592
Statistical Analysis 1: Comparison: Rayaldee vs Placebo; Test type: Other; p = 0.7856, Regression, Logistic; Logistic regression with treatment as the main effect, and baseline aggregate symptom score, baseline 25D level, and body weight as covariates

6. Secondary Outcome: Number of Participants With Emergency Room/Urgent Care Visits
Description: Number and percentage of subjects with emergency room/urgent care visits
Time Frame: 42 days
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Rayaldee | Placebo
Number analyzed (Participants) | 65 | 69
Participants | 0 | 3

7. Secondary Outcome: Number of Participants With Oxygen Saturation Below 94% (Without Supplemental Oxygen)
Description: Number and percentage of subjects with oxygen saturation below 94% (without supplemental oxygen)
Time Frame: 42 days
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Rayaldee | Placebo
Number analyzed (Participants) | 65 | 69
Participants | 0 | 1

8. Secondary Outcome: Number of Participants With Hospitalizations
Description: Number and percentage of subjects with hospitalization
Time Frame: 42 days
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Rayaldee | Placebo
Number analyzed (Participants) | 65 | 69
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With the Requirement for Mechanical Ventilation
Description: Number and percentage of subjects requiring mechanical ventilation
Time Frame: 42 days
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Rayaldee | Placebo
Number analyzed (Participants) | 65 | 69
Participants | 0 | 0

10. Secondary Outcome: Number of Participant Deaths
Description: Number and percentage of subjects who died
Time Frame: 42 days
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Rayaldee | Placebo
Number analyzed (Participants) | 65 | 69
Participants | 0 | 0

11. Secondary Outcome: Severity of COVID-19 Illness as Evidenced by Quality of Life Measures Using the FLU-PRO Plus Questionnaire
Description: Quality-of-Life (QOL) responses are based on the number of non-missing observations within individual QOL question and visit. Comparisons to baseline are assessed only for subjects who were at risk for improvement. Percentages for the comparisons to baseline are based on the number at-risk for improvement.
Time Frame: 14 days
Population: Per protocol population at-risk for improvement from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Rayaldee | Placebo
Number analyzed (Participants) | 65 | 69
Participants
  Overall, how severe were your infection symptoms today?: number analyzed (Participants) | 65 | 66
  Overall, how severe were your infection symptoms today?: Improved compared to baseline | 47 | 48
  Overall, how severe were your infection symptoms today?: Worsened compared to baseline | 1 | 1
  Overall, how severe were your infection symptoms today?: No charge from baseline | 5 | 7
  Overall, how severe were your infection symptoms today?: Missing | 12 | 10
  Overall, how were your infection symptoms today compared to yesterday?: number analyzed (Participants) | 65 | 68
  Overall, how were your infection symptoms today compared to yesterday?: Improved compared to baseline | 45 | 50
  Overall, how were your infection symptoms today compared to yesterday?: Worsened compared to baseline | 0 | 1
  Overall, how were your infection symptoms today compared to yesterday?: No charge from baseline | 8 | 7
  Overall, how were your infection symptoms today compared to yesterday?: Missing | 12 | 10
  How much did your infection symptoms interfere with your usual activities today?: number analyzed (Participants) | 65 | 67
  How much did your infection symptoms interfere with your usual activities today?: Improved compared to baseline | 48 | 52
  How much did your infection symptoms interfere with your usual activities today?: Worsened compared to baseline | 1 | 0
  How much did your infection symptoms interfere with your usual activities today?: No charge from baseline | 4 | 5
  How much did your infection symptoms interfere with your usual activities today?: Missing | 12 | 10
  Have you returned to your usual activities today?: number analyzed (Participants) | 64 | 68
  Have you returned to your usual activities today?: Improved compared to baseline | 26 | 34
  Have you returned to your usual activities today?: Worsened compared to baseline | 0 | 0
  Have you returned to your usual activities today?: No charge from baseline | 26 | 24
  Have you returned to your usual activities today?: Missing | 12 | 10
  In general, how would you rate your physical health today?: Improved compared to baseline | 48 | 47
  In general, how would you rate your physical health today?: Worsened compared to baseline | 0 | 1
  In general, how would you rate your physical health today?: No charge from baseline | 5 | 10
  In general, how would you rate your physical health today?: Missing | 12 | 11
  Have you returned to your usual health today?: number analyzed (Participants) | 65 | 68
  Have you returned to your usual health today?: Improved compared to baseline | 19 | 19
  Have you returned to your usual health today?: Worsened compared to baseline | 0 | 0
  Have you returned to your usual health today?: No charge from baseline | 34 | 39
  Have you returned to your usual health today?: Missing | 12 | 10

12. Secondary Outcome: Resolution of Symptoms Based on FLU-PRO Plus© COVID-19 Five Symptom Aggregate Score Based on Serum 25D Level Over the Treatment Period
Description: Clinical course of COVID-19 as a function of Serum Total 25-hydroxyvitamin D concentrations of <50 ng/mL, 50 to 100 ng/mL and >100 ng/mL at Day 14, defined as the proportion of subjects in each treatment group with a total score of ≤5 for the selected five COVID-19 symptoms (trouble breathing, chest congestion, dry or hacking cough, body aches and pains, and chills and shivering) using the FLU-PRO Plus© questionnaire. Results were similar for comparisons between treatment groups on Days 7, 14, 21 and 28, and only data for Day 14 is presented.
Time Frame: 14 days
Population: Per protocol population minus the number of participants with missing observations (4 participants in each Arm/Group).
Measure: Count of Participants; unit: Participants
Arm/Group | Rayaldee | Placebo
Number analyzed (Participants) | 61 | 65
Participants
  Serum 25D Level <50 ng/mL: number analyzed (Participants) | 10 | 55
  Serum 25D Level <50 ng/mL: Yes | 4 | 38
  Serum 25D Level <50 ng/mL: No | 6 | 17
  Serum 25D Level 50 - 100 ng/mL: number analyzed (Participants) | 36 | 10
  Serum 25D Level 50 - 100 ng/mL: Yes | 28 | 8
  Serum 25D Level 50 - 100 ng/mL: No | 8 | 2
  Serum 25D Level >100 ng/mL: number analyzed (Participants) | 15 | 0
  Serum 25D Level >100 ng/mL: Yes | 11 | 0
  Serum 25D Level >100 ng/mL: No | 4 | 0

ADVERSE EVENTS:
Time Frame: 42 days
Description: Analysis is for the safety population, subjects who received any amount of study drug treatment.
Arm/Group | Rayaldee | Placebo
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 3/80 | 1/80
Other Adverse Events (participants affected / at risk) | 12/80 | 12/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rayaldee (N=80) | Placebo (N=80)
COVID-19 pneumonia (Infections and infestations) | 3 | 0
COVID-19 (Infections and infestations) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rayaldee (N=80) | Placebo (N=80)
COVID-19 (Infections and infestations) | 0 | 5
COVID-19 pneumonia (Infections and infestations) | 3 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Electrocardiogram ST-T segment abnormal (Investigations) | 1 | 1
Transaminases increased (Investigations) | 2 | 0
Blood parathyroid hormone increased (Investigations) | 1 | 0
Blood sodium decreased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 0
Electrocardiogram QRS complex abnormal (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
A caveat in the analysis is the variability of 25D at baseline. The study is also limited by timing differences between the onset of symptoms and diagnosis of COVID-19, and between COVID-19 diagnosis and the initiation of treatment among participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT04551911/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT04551911/SAP_001.pdf